CLINICAL TRIAL: NCT04835597
Title: Precision Performance Status Assessment in Breast Cancer Patients Receiving Neoadjuvant Chemotherapy
Status: Terminated | Type: Observational
Why Stopped: IRB Study Closure
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1237; NCI-2021-02624 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1237 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (movement assessment, medical data collection): Patients complete movement assessment 5-15 days prior to the initiation of neoadjuvant chemotherapy and at day 1 of neoadjuvant chemotherapy. Patients' SAE data is collected. Patients are observed during their neoadjuvant chemotherapy for up to 6 months.
  Interventions: Behavioral: Behavioral Assessment; Other: Electronic Health Record Review

INTERVENTIONS:
Behavioral: Behavioral Assessment — Complete movement assessment
Other: Electronic Health Record Review — SAE data is collected

SUMMARY:
This study assesses the performance status in stage I-III triple negative breast cancer patients who are receiving neoadjuvant chemotherapy. Information collected in this study may help doctors learn if movement and fitness trackers can be used to predict side effects in cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if in-office movement trackers or baseline metabolic equivalents (METs) groups identify those patients who are at highest risk for severe adverse event (SAE)s on neoadjuvant chemotherapy.

SECONDARY OBJECTIVES:

I. To determine the association between the occurrence of SAEs, unexpected healthcare encounters, depending on the change in activity level classification between the baseline METs group and mid-treatment METs group (at month 3).

II. Explore association between patient reported outcome (PRO) data and movement tracker data.

OUTLINE:

Patients complete movement assessment 5-15 days prior to the initiation of neoadjuvant chemotherapy and at day 1 of neoadjuvant chemotherapy. Patients' SAE data is collected. Patients are observed during their neoadjuvant chemotherapy for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed breast cancer with any receptor status, who will receive neoadjuvant chemotherapy. Patients with denovo oligo-metastatic disease, where the intent of therapy is curative with incorporation of local therapy (surgery/radiation to the breast and/or metastatic sites) are also eligible.
* Age >= 18 years
* Ability to understand and the willingness to sign a written informed consent
* Willingness to wear sensors to track physical activity, global positioning system (GPS) location, and provide symptom ratings each night during the screening period of their clinical trial and 180 days after starting treatments
* Able to read English, Spanish, or Mandarin to complete patient reported outcomes
* Able to ambulate without an assistive device

Exclusion Criteria:

* Missing lower limbs
* Known movement disorder such as Parkinson's disease, choreo-athetoid movement disorders, essential tremor if that movement disorder is of sufficient severity to require drug therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with triple negative breast cancer who will receive neoadjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
The number of non-hematologic serious adverse events occurring during neoadjuvant chemotherapy (i.e. correlate Microsoft motion tracking data and baseline metabolic equivalents [METs] group with incidence of serious adverse events) | Up to 6 months

SECONDARY OUTCOMES:
The number of severe adverse event (SAE)s | During the final 3 months of neoadjuvant chemotherapy
The number of SAEs based on laboratory results | Over the final 3 months of neoadjuvant chemotherapy
The number of SAEs based on symptoms | Over the final 3 months of neoadjuvant chemotherapy
The number of unexpected healthcare encounters | In the final 3 months of neoadjuvant chemotherapy
Correlation between patient reported outcomes (PRO) data and movement tracker data | 6 months
  Will calculate the Pearson correlation between PRO data and movement tracker data. Will also fit a linear mixed model with PRO data as the dependent variable and movement tracker data as covariates. Intra-subject correlation will be adjusted in linear mixed model analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Karuturi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org